CLINICAL TRIAL: NCT04013412
Title: Dietary Restriction in Vascular Surgery
Acronym: DRIVeS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, C. Keith Ozaki, M.D., F.A.C.S., John A. Mannick Professor of Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018P002133
Record Dates: First submitted 2019-06-24; First posted 2019-07-09 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Vascular Diseases; Surgery
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: 3:2 randomization to short-term protein calorie restriction diet versus regular meals prior to elective major vascular surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-Calorie Restriction (Experimental): Four day dietary intervention immediately before surgery of ScandiShake [any of 4 flavors] mixed with almond milk, calculated individually for a total daily volume to achieve 30% caloric restriction and 70% protein restriction, based on body weight and activity level.
  Interventions: Dietary Supplement: Protein-Calorie Restriction
- Control (No Intervention): Ad libitum diet for four days immediately before surgery

INTERVENTIONS:
Dietary Supplement: Protein-Calorie Restriction — Four day dietary intervention immediately before surgery of ScandiShake [any of 4 flavors] mixed with almond milk, calculated individually for a total daily volume to achieve 30% caloric restriction and 70% protein restriction, based on body weight and activity level.
  Arms: Protein-Calorie Restriction

SUMMARY:
A randomized, controlled trial to evaluate patient compliance and biologic mechanisms of a short-term pre-operative Protein-Calorie Restriction (PCR) diet in comparison to a normal ad libitum diet for 4 days before elective vascular surgery involving a major operation. This study is a step in the long-term primary scientific objective to test the hypothesis that brief up regulation of endogenous H2S via pre-operative PCR in elective major surgery improves clinical outcomes in humans. After a successful pilot study of the PCR diet conducted inpatient before carotid endarterectomy, the investigators now aim to expand the study to at home diet among a variety of vascular surgery procedures.

DETAILED DESCRIPTION:
Hydrogen sulfide (H2S) has emerged as a critical gaseous signaling molecule with a role in multiple processes including ischemia-reperfusion (IR) injury, angiogenesis, intimal hyperplasia, and anti-inflammatory mechanisms. It even appears to hold anti-atherosclerotic properties. However, the gas is toxic with a half-life of minutes, and it can be rapidly oxidized. Furthermore, no clinically useful pharmacologic H2S donors have been developed to date. In a 2015 Cell paper, the study investigators link substantial upregulation of endogenous H2S to short-term manipulation of mammalian dietary intake: simple dietary restriction. The current project serves as the second phase in the accelerated translation of this important discovery toward clinical utility that may substantively impact the vascular patient at several levels: protection from IR injury, intimal hyperplasia, peri-procedural events such as stroke, cardiac dysfunction and myocardial infarction (MI), and promotion of angiogenesis.

Chronic protein and calorie dietary restriction (PCR; reduced food intake without malnutrition) is known for extending longevity in multiple species. PCR is also an established approach to positively impact metabolic fitness and resistance to multiple forms of acute stress. Despite these wide-ranging benefits, potential clinical applications have never been considered feasible in humans due to the practical difficulties associated with voluntary food restriction combined with the assumption that PCR benefits take a long time to accrue. Recent preclinical studies by the applicants reveal a rapid onset of PCR benefits against surgically induced traumatic inflammation, IR injury, and the fibroproliferative vascular response to injury in rodents. Mechanistically, rapid changes in adipose phenotype and associated adipokine profiles appear to underlie these benefits; but the key mediator appears to be endogenous H2S. This field thus stands poised to move to clinical utility, and vascular surgery offers an optimal risk/benefit ratio for translation of the PCR/H2S hypothesis.

For the current project the investigators will complete a randomized, controlled trial to evaluate patient compliance and biologic mechanisms of a short-term pre-operative PCR diet in comparison to a normal ad libitum diet for 4 days before elective major vascular surgery. Both Endpoints relate to the long-term primary scientific objective to test the hypothesis that brief upregulation of endogenous H2S via pre-operative PCR in elective major surgery improves clinical outcomes in humans. After a successful pilot study of the PCR diet conducted inpatient before carotid endarterectomy titled Short-Term Endogenous Hydrogen Sulfide Upregulation (NCT03303534), the investigators now aim to expand the study to at home diet among a variety of vascular surgery procedures.

Eighty subjects undergoing carotid artery endarterectomy, aortic aneurysm repair (open, and endovascular if groin cut down planned), open lower extremity arterial procedures (bypasses, aneurysm repair, arterial and bypass graft reconstructions), major amputation of the lower extremity (below knee and above knee amputations), or open hemodialysis access procedures for either symptomatic or asymptomatic disease will be recruited and enrolled at Brigham and Women's Hospital. Using a randomized (3:2), parallel design, patients will receive either the PCR diet (n=48; ScandiShake [any of 4 flavors] mixed with almond milk, calculated individually for a total daily volume to achieve 30% caloric restriction and 70% protein restriction, based on body weight and activity level), or continued routine ad libitum diet (n=32). Daily physical activity will be assessed by questionnaire to determine the activity factor for accurate calorie restriction calculations. Water intake is ad libitum for both cohorts, and both diets can be consumed throughout the day and night (except on the day of surgery). Patients will consume their assigned diets for the four days leading up to surgery until midnight the day of surgery when both cohorts will be fasted for the procedure (per standard clinical guidelines).

ELIGIBILITY:
Inclusion Criteria

• Patients greater than 18 years old who present for one of the following elective procedures at Brigham and Women's Hospital

* Carotid artery endarterectomy
* Aortic/iliac aneurysm repair (open, and endovascular if groin cut down planned)
* Open lower extremity arterial procedures (bypasses, aneurysm repair, arterial and bypass graft reconstructions)
* Major amputation of the lower extremity (below knee and above knee amputations).
* Open hemodialysis access procedures

Exclusion Criteria

* Patient intolerance or allergy to any of the ingredients in the PCR diet
* Active infection
* Pregnancy
* Malnutrition, based on abnormally low serum albumin (lower than 3 g/dL)
* Uncontrolled diabetes (HgbA1c greater than 12%)
* Substance dependency that could interfere with protocol adherence and assent as determined by the PI
* Active non-cutaneous cancer under treatment with chemotherapeutics or radiation
* Emergency surgery
* Active participation in any another interventional or randomized study
* Participation in the current study within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Outpatient compliance with protein calorie restriction | 1 Month
  Patient compliance with the PCR diet will be assessed by food record analysis.
Comparison of H2S and related biological markers of stress | 1 Month
  Biologic markers include: adipose phenotyping (quantification of adipokines, adipose derived hormones), leukocyte phenotyping and quantification via flow cytometry, and serum assays of IL-1beta, IL-6, IL-8, HGF, leptin, MCP-1, PAI-1, resistin, NGF, TNF, adiponectin, hydrogen sulfide (including production capacity) assays, insulin, lipid panels, FGF 21, pre-albumin, epinephrine, norepinephrine, dopamine, CBC with differential, basic metabolic panel including calcium. H2S and biologic markers will be compared at baseline, immediately before surgery, and the day after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Charles K Ozaki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hine C, Kim HJ, Zhu Y, Harputlugil E, Longchamp A, Matos MS, Ramadoss P, Bauerle K, Brace L, Asara JM, Ozaki CK, Cheng SY, Singha S, Ahn KH, Kimmelman A, Fisher FM, Pissios P, Withers DJ, Selman C, Wang R, Yen K, Longo VD, Cohen P, Bartke A, Kopchick JJ, Miller R, Hollenberg AN, Mitchell JR. Hypothalamic-Pituitary Axis Regulates Hydrogen Sulfide Production. Cell Metab. 2017 Jun 6;25(6):1320-1333.e5. doi: 10.1016/j.cmet.2017.05.003. PMID 28591635
- [Background] Longchamp A, Harputlugil E, Corpataux JM, Ozaki CK, Mitchell JR. Is Overnight Fasting before Surgery Too Much or Not Enough? How Basic Aging Research Can Guide Preoperative Nutritional Recommendations to Improve Surgical Outcomes: A Mini-Review. Gerontology. 2017;63(3):228-237. doi: 10.1159/000453109. Epub 2017 Jan 5. PMID 28052287
- [Background] Longchamp A, Tao M, Bartelt A, Ding K, Lynch L, Hine C, Corpataux JM, Kristal BS, Mitchell JR, Ozaki CK. Surgical injury induces local and distant adipose tissue browning. Adipocyte. 2015 Nov 20;5(2):163-74. doi: 10.1080/21623945.2015.1111971. eCollection 2016 Apr-Jun. PMID 27386152
- [Background] Robertson LT, Trevino-Villarreal JH, Mejia P, Grondin Y, Harputlugil E, Hine C, Vargas D, Zheng H, Ozaki CK, Kristal BS, Simpson SJ, Mitchell JR. Protein and Calorie Restriction Contribute Additively to Protection from Renal Ischemia Reperfusion Injury Partly via Leptin Reduction in Male Mice. J Nutr. 2015 Aug;145(8):1717-27. doi: 10.3945/jn.114.199380. Epub 2015 Jun 3. PMID 26041674
- [Background] Hine C, Harputlugil E, Zhang Y, Ruckenstuhl C, Lee BC, Brace L, Longchamp A, Trevino-Villarreal JH, Mejia P, Ozaki CK, Wang R, Gladyshev VN, Madeo F, Mair WB, Mitchell JR. Endogenous hydrogen sulfide production is essential for dietary restriction benefits. Cell. 2015 Jan 15;160(1-2):132-44. doi: 10.1016/j.cell.2014.11.048. Epub 2014 Dec 23. PMID 25542313
- [Background] Mauro CR, Tao M, Yu P, Trevino-Villerreal JH, Longchamp A, Kristal BS, Ozaki CK, Mitchell JR. Preoperative dietary restriction reduces intimal hyperplasia and protects from ischemia-reperfusion injury. J Vasc Surg. 2016 Feb;63(2):500-9.e1. doi: 10.1016/j.jvs.2014.07.004. Epub 2014 Aug 8. PMID 25124359
- [Background] Nguyen B, Tao M, Yu P, Mauro C, Seidman MA, Wang YE, Mitchell J, Ozaki CK. Preoperative diet impacts the adipose tissue response to surgical trauma. Surgery. 2013 Apr;153(4):584-93. doi: 10.1016/j.surg.2012.11.001. Epub 2012 Dec 27. PMID 23274098
- [Background] Mitchell JR, Beckman JA, Nguyen LL, Ozaki CK. Reducing elective vascular surgery perioperative risk with brief preoperative dietary restriction. Surgery. 2013 Apr;153(4):594-8. doi: 10.1016/j.surg.2012.09.007. Epub 2012 Dec 4. PMID 23218877

DOCUMENTS (2):
  • Informed Consent Form (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT04013412/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04013412/Prot_SAP_001.pdf